CLINICAL TRIAL: NCT07207603
Title: Observational Cohort Pilot Study on Cardiovascular Prevention in Citizens Living in Milano-Bicocca District
Brief Title: Bicocca Epidemiological Assessment of Cardiovascular Risk Factors
Acronym: MUSA-BEA
Status: Enrolling by invitation | Type: Observational
Sponsor: University of Milano Bicocca (Other)
Collaborators: Istituto Auxologico Italiano (Other)
Responsible Party: Sponsor
Other Study IDs: BEA 777
Record Dates: First submitted 2024-09-20; First posted 2025-10-06 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-10

CONDITIONS: Cardiovascular Risk Factors (e.g., Hypertension)
Keywords: Cardiovascular risk factor; Italy; Observational Study; Epidemiology; exposome; air pollution; blood pressure; cholesterol; stress
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Bloods will be taken by a dedicated Research Nurse and sent for analysis and storage. In detail 5 vacutainers (5 ml each) will be taken for each subject and the following analyses will be performed: glucose level, total cholesterol, HDL, triglycerides, LDLc, ApoB, Lp(a), HbA1c, uric acid, hsPCR. Urine samples will be also collected for urine analysis. Furthermore, two 80 mg stool aliquots will be stored allowing the possibility of evaluating the gut microbiome composition.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Recruited individuals: Males or females age > 25 years living in the area close to University Milano-Bicocca (postcode 20126) and able to sign the informed consent.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
The main objective of the study is to characterize the cardiovascular risk profile of the population in the Bicocca district through the evaluation of the exposome and the assessment of traditional and less studied cardiovascular risk factors for cardiovascular disease.

DETAILED DESCRIPTION:
STUDY DURATION AND ENROLMENT

The study duration is 3 years. The study will be conducted at University of Milano-Bicocca in an ad-hoc site dedicated to the project.

STUDY POPULATION

Inclusion Criteria: Males or females age > 25 years living in the area close to University Milano-Bicocca (postcode 20126) Exclusion Criteria: Inability to sign the informed consent

STUDY PROCEDURES During the screening visit the Investigators will double check that the subject can be included according to the aforementioned inclusion and exclusion criteria.

Informed Consent will be signed by both Investigator and Subject enrolled.

OBSERVATIONAL PERIOD

If the screening visit is successful (if the subjects meet the inclusion criteria and does not meet the exclusion criteria) the main visit will be scheduled or can be performed at the same time of the screening visit if feasible. If possible, all study procedures will be performed on the same day. If not, the study procedures will be scheduled and the subject will be invited to come in the following days. If possible, self-report questionnaires not requiring any supervision will be administered digitally through an ad hoc web platform (i.e., Qualtrics) in order to save time and reduce the participant's time spent at the research facility.

STUDY EVALUATIONS AND MEASUREMENTS

* Demographic and clinical characteristics;
* Medical history;
* Current treatment;
* Physiscal examination;
* Vital signs;
* Laboratory evaluations;
* Questionaires (lifestyle profiles; cognitive functions; psychological dispositions; health-related psychological dispositions; perceived health and wellbeing; stress);
* Frailty assessment (in elderly participants only)
* Lung Function test;
* ECG/Ambulatory blood pressure measurement/heandgrip test/PWA and PWV assessment/optical cohoerence tomography angiography and non-mydriatic fundus retinography/Air pollutant assessment

STATISTICAL ANALYSIS Data will be summarised by standard descriptive summaries (e.g. means and standard deviations for continuous variables such as age and percentages for categorical variables such as gender). Appropriate statistical methods will be adopted to assess the association between cardiovascular factors and global cardiovascular risk profile.

ELIGIBILITY:
Inclusion Criteria:

* Individuals living in the area close to University Milano-Bicocca (postcode 20126)

Exclusion Criteria:

* Inability to sign the informed consent

Min Age: 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Our target population includes about 15900 residents in the 20126 postcode area with at least 25 years of age. From this population we aim to select a sample of 1000 subjects which will participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-06-17 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Exposome | prior index date and at baseline visit
  to define the prevalence of the exposome associated with increased CV risk in an urban population.
  The exposome includes the following domains:
  1. Internal: internal biological processes such as oxidative stress, inflammation, epigenetic changes, metabolism and the internal microbiome.
  2. General external: social, economic factors, the urban environment and climate factors.
  3. Specific external: an individual's immediate local environment, including exposure to chemicals, diet, physical activity, tobacco and infections.

SECONDARY OUTCOMES:
Traditional CV risk factors | prior index date and at baseline visit
  the prevalence of the known CV risk factors (e.g., high blood pressure, diabetes, smoking status, dyslipidaemia) will be evaluated according to current Guidelines for Cardiovascular Prevention.
  In addition to this the following known risk factors will be determined as follows
  * The non-adequacy of physical activity will be established based on the IPAQ total score. A score below 3000 MET-minute/week is indicative of an inactive lifestyle. Also, the categorical score that identifies "inactive," "minimally active," and "HEPA active" will be used to classify participants;
  * The non-adequacy of eating habits will be established based on the MD score of the QueMD scale. A score below 5 suggests good adherence to the Mediterranean diet;
  * Alcohol consumption will be evaluated through the individual scores on the AUDIT-C. A score equal to or greater than 5 for males and equal to or greater than 4 for females indicates a possible risky consumption of alcohol.
Non traditional risk factors | prior index date and at baseline visit
  prevalence of new/less studied risk modifiers (including psychological profiles associated with unhealthy lifestyle and misperception of CV risk) in an urban population.
  Specifically:
  * the prevalence of psychosocial stress will be determined through the evaluation of individual scores on the PSS.
  * the presence of anxiety symptoms will be determined by evaluating individual scores on the GAD-7;
  * the presence of depressive symptoms will be evaluated through the individual scores on the PHQ-9;
  * the prevalence of frailty in the elderly participants will be determined according to the Fried's frailty phenotype;
  * the prevalence of short (<6 hours of sleep) and long sleepers (>8 hours of sleep) will be defined by the Pittsburgh sleep quality index;
  * the prevalence of low socioeconomic status will be determined as well as work stress defined by job strain (i.e. the combination of high demands and low control at work) and effort-reward imbalance.

OTHER OUTCOMES:
Prevalence of clinical conditions associated with CV risk | prior index date and at baseline visit
  The prevalence of clinical conditions associated with CV risk will be determined as follows:
  * The prevalence of sleep disturbances will be defined according to the presence of sleep disorders as defined by the International Classification of Sleep Disorders (third edition);
  * The prevalence of cancer will be determined based on past medical history;
  * The prevalence of chronic obstructive pulmonary disease will be determined based on past medical history and will be supported by the results of spirometry;
  * The prevalence of migraine will be determined based on past medical history;
  * The prevalence of erectile dysfunction, defined as the consistent inability to reach and maintain an erection satisfactory for sexual activity will be determined based on past medical history
  * The prevalence of polycystic ovary syndrome and premature menopause will be determined based on past medical history
  * The prevalence of inflammatory conditions such as rheumatoid arthritis, psoriasis and ankylos

CONTACTS AND LOCATIONS:
Overall Officials: Martino F Pengo, Medicine, Principal Investigator — University of Milan-Bicocca
Locations (1):
- University of Milan-Bicocca, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Luciani M, De Maria M, Page SD, Barbaranelli C, Ausili D, Riegel B. Measuring self-care in the general adult population: development and psychometric testing of the Self-Care Inventory. BMC Public Health. 2022 Mar 28;22(1):598. doi: 10.1186/s12889-022-12913-7. PMID 35346104
- [Result] Chang VT, Hwang SS, Feuerman M, Kasimis BS, Thaler HT. The memorial symptom assessment scale short form (MSAS-SF). Cancer. 2000 Sep 1;89(5):1162-71. doi: 10.1002/1097-0142(20000901)89:53.0.co;2-y. PMID 10964347
- [Result] Cali G, Ambrosini E, Picconi L, Mehling WE, Committeri G. Investigating the relationship between interoceptive accuracy, interoceptive awareness, and emotional susceptibility. Front Psychol. 2015 Aug 24;6:1202. doi: 10.3389/fpsyg.2015.01202. eCollection 2015. PMID 26379571
- [Result] Schandry R. Heart beat perception and emotional experience. Psychophysiology. 1981 Jul;18(4):483-8. doi: 10.1111/j.1469-8986.1981.tb02486.x. No abstract available. PMID 7267933
- [Result] Kontiola A. A new electromechanical method for measuring intraocular pressure. Doc Ophthalmol. 1996-1997;93(3):265-76. doi: 10.1007/BF02569066. PMID 9550354
- [Result] Curcio G, Tempesta D, Scarlata S, Marzano C, Moroni F, Rossini PM, Ferrara M, De Gennaro L. Validity of the Italian version of the Pittsburgh Sleep Quality Index (PSQI). Neurol Sci. 2013 Apr;34(4):511-9. doi: 10.1007/s10072-012-1085-y. Epub 2012 Apr 13. PMID 22526760
- [Result] Picardi A, Adler DA, Abeni D, Chang H, Pasquini P, Rogers WH, Bungay KM. Screening for depressive disorders in patients with skin diseases: a comparison of three screeners. Acta Derm Venereol. 2005;85(5):414-9. doi: 10.1080/00015550510034966. PMID 16159733
- [Result] Lorini C, Lastrucci V, Mantwill S, Vettori V, Bonaccorsi G; Florence Health Literacy Research Group. Measuring health literacy in Italy: a validation study of the HLS-EU-Q16 and of the HLS-EU-Q6 in Italian language, conducted in Florence and its surroundings. Ann Ist Super Sanita. 2019 Jan-Mar;55(1):10-18. doi: 10.4415/ANN_19_01_04. PMID 30968831
- [Result] Steca P, Monzani D, Pierobon A, Avvenuti G, Greco A, Giardini A. Measuring dispositional optimism in patients with chronic heart failure and their healthcare providers: the validity of the Life Orientation Test-Revised. Patient Prefer Adherence. 2017 Sep 6;11:1497-1503. doi: 10.2147/PPA.S139522. eCollection 2017. PMID 28919722
- [Result] Poreh A, Bezdicek O, Korobkova I, Levin JB, Dines P. The Rey Auditory Verbal Learning Test forced-choice recognition task: Base-rate data and norms. Appl Neuropsychol Adult. 2016;23(3):155-61. doi: 10.1080/23279095.2015.1027343. Epub 2015 Oct 27. PMID 26507316
- [Result] Rekers S, Finke C. Translating spatial navigation evaluation from experimental to clinical settings: The virtual environments navigation assessment (VIENNA). Behav Res Methods. 2024 Mar;56(3):2033-2048. doi: 10.3758/s13428-023-02134-0. Epub 2023 May 11. PMID 37166580
- [Result] Ragland JD, Turetsky BI, Gur RC, Gunning-Dixon F, Turner T, Schroeder L, Chan R, Gur RE. Working memory for complex figures: an fMRI comparison of letter and fractal n-back tasks. Neuropsychology. 2002 Jul;16(3):370-9. PMID 12146684
- [Result] Morisky DE, Green LW, Levine DM. Concurrent and predictive validity of a self-reported measure of medication adherence. Med Care. 1986 Jan;24(1):67-74. doi: 10.1097/00005650-198601000-00007. PMID 3945130
- [Result] Adorni R, Zanatta F, D'Addario M, Atella F, Costantino E, Iaderosa C, Petarle G, Steca P. Health-Related Lifestyle Profiles in Healthy Adults: Associations with Sociodemographic Indicators, Dispositional Optimism, and Sense of Coherence. Nutrients. 2021 Oct 25;13(11):3778. doi: 10.3390/nu13113778. PMID 34836035
- [Result] Gnagnarella P, Draga D, Misotti AM, Sieri S, Spaggiari L, Cassano E, Baldini F, Soldati L, Maisonneuve P. Validation of a short questionnaire to record adherence to the Mediterranean diet: An Italian experience. Nutr Metab Cardiovasc Dis. 2018 Nov;28(11):1140-1147. doi: 10.1016/j.numecd.2018.06.006. Epub 2018 Jun 18. PMID 30077491
- [Result] Choi M, Mesa-Frias M, Nuesch E, Hargreaves J, Prieto-Merino D, Bowling A, Snith GD, Ebrahim S, Dale C, Casas JP. Social capital, mortality, cardiovascular events and cancer: a systematic review of prospective studies. Int J Epidemiol. 2014 Dec;43(6):1895-920. doi: 10.1093/ije/dyu212. PMID 25369975
- [Result] Parati G, Stergiou GS, Bilo G, Kollias A, Pengo M, Ochoa JE, Agarwal R, Asayama K, Asmar R, Burnier M, De La Sierra A, Giannattasio C, Gosse P, Head G, Hoshide S, Imai Y, Kario K, Li Y, Manios E, Mant J, McManus RJ, Mengden T, Mihailidou AS, Muntner P, Myers M, Niiranen T, Ntineri A, O'Brien E, Octavio JA, Ohkubo T, Omboni S, Padfield P, Palatini P, Pellegrini D, Postel-Vinay N, Ramirez AJ, Sharman JE, Shennan A, Silva E, Topouchian J, Torlasco C, Wang JG, Weber MA, Whelton PK, White WB, Mancia G; Working Group on Blood Pressure Monitoring and Cardiovascular Variability of the European Society of Hypertension. Home blood pressure monitoring: methodology, clinical relevance and practical application: a 2021 position paper by the Working Group on Blood Pressure Monitoring and Cardiovascular Variability of the European Society of Hypertension. J Hypertens. 2021 Sep 1;39(9):1742-1767. doi: 10.1097/HJH.0000000000002922. PMID 34269334
- [Result] Williams B, Mancia G, Spiering W, Agabiti Rosei E, Azizi M, Burnier M, Clement DL, Coca A, de Simone G, Dominiczak A, Kahan T, Mahfoud F, Redon J, Ruilope L, Zanchetti A, Kerins M, Kjeldsen SE, Kreutz R, Laurent S, Lip GYH, McManus R, Narkiewicz K, Ruschitzka F, Schmieder RE, Shlyakhto E, Tsioufis C, Aboyans V, Desormais I; Authors/Task Force Members:. 2018 ESC/ESH Guidelines for the management of arterial hypertension: The Task Force for the management of arterial hypertension of the European Society of Cardiology and the European Society of Hypertension: The Task Force for the management of arterial hypertension of the European Society of Cardiology and the European Society of Hypertension. J Hypertens. 2018 Oct;36(10):1953-2041. doi: 10.1097/HJH.0000000000001940. PMID 30234752
- [Result] Ikram MA, Brusselle GGO, Murad SD, van Duijn CM, Franco OH, Goedegebure A, Klaver CCW, Nijsten TEC, Peeters RP, Stricker BH, Tiemeier H, Uitterlinden AG, Vernooij MW, Hofman A. The Rotterdam Study: 2018 update on objectives, design and main results. Eur J Epidemiol. 2017 Sep;32(9):807-850. doi: 10.1007/s10654-017-0321-4. Epub 2017 Oct 24. PMID 29064009
- [Result] Brodaty H, Pond D, Kemp NM, Luscombe G, Harding L, Berman K, Huppert FA. The GPCOG: a new screening test for dementia designed for general practice. J Am Geriatr Soc. 2002 Mar;50(3):530-4. doi: 10.1046/j.1532-5415.2002.50122.x. PMID 11943052
- [Result] Galvin JE, Roe CM, Powlishta KK, Coats MA, Muich SJ, Grant E, Miller JP, Storandt M, Morris JC. The AD8: a brief informant interview to detect dementia. Neurology. 2005 Aug 23;65(4):559-64. doi: 10.1212/01.wnl.0000172958.95282.2a. PMID 16116116
- [Result] Guralnik JM, Ferrucci L, Pieper CF, Leveille SG, Markides KS, Ostir GV, Studenski S, Berkman LF, Wallace RB. Lower extremity function and subsequent disability: consistency across studies, predictive models, and value of gait speed alone compared with the short physical performance battery. J Gerontol A Biol Sci Med Sci. 2000 Apr;55(4):M221-31. doi: 10.1093/gerona/55.4.m221. PMID 10811152
- [Result] Di Castelnuovo A, Costanzo S, Persichillo M, Olivieri M, de Curtis A, Zito F, Donati MB, de Gaetano G, Iacoviello L; MOLI-SANI Project Investigators. Distribution of short and lifetime risks for cardiovascular disease in Italians. Eur J Prev Cardiol. 2012 Aug;19(4):723-30. doi: 10.1177/1741826711410820. Epub 2011 May 13. PMID 21571772
- [Result] Farooqi MAM, Gerstein H, Yusuf S, Leong DP. Accumulation of Deficits as a Key Risk Factor for Cardiovascular Morbidity and Mortality: A Pooled Analysis of 154 000 Individuals. J Am Heart Assoc. 2020 Feb 4;9(3):e014686. doi: 10.1161/JAHA.119.014686. Epub 2020 Jan 28. PMID 31986990
- [Result] Purser JL, Kuchibhatla MN, Fillenbaum GG, Harding T, Peterson ED, Alexander KP. Identifying frailty in hospitalized older adults with significant coronary artery disease. J Am Geriatr Soc. 2006 Nov;54(11):1674-81. doi: 10.1111/j.1532-5415.2006.00914.x. PMID 17087693
- [Result] Iwasaki A, Pillai PS. Innate immunity to influenza virus infection. Nat Rev Immunol. 2014 May;14(5):315-28. doi: 10.1038/nri3665. PMID 24762827
- [Result] Munzel T, Sorensen M, Hahad O, Nieuwenhuijsen M, Daiber A. The contribution of the exposome to the burden of cardiovascular disease. Nat Rev Cardiol. 2023 Oct;20(10):651-669. doi: 10.1038/s41569-023-00873-3. Epub 2023 May 10. PMID 37165157
- [Result] Visseren FLJ, Mach F, Smulders YM, Carballo D, Koskinas KC, Back M, Benetos A, Biffi A, Boavida JM, Capodanno D, Cosyns B, Crawford C, Davos CH, Desormais I, Di Angelantonio E, Franco OH, Halvorsen S, Hobbs FDR, Hollander M, Jankowska EA, Michal M, Sacco S, Sattar N, Tokgozoglu L, Tonstad S, Tsioufis KP, van Dis I, van Gelder IC, Wanner C, Williams B; ESC National Cardiac Societies; ESC Scientific Document Group. 2021 ESC Guidelines on cardiovascular disease prevention in clinical practice. Eur Heart J. 2021 Sep 7;42(34):3227-3337. doi: 10.1093/eurheartj/ehab484. No abstract available. PMID 34458905
- See also: Related Info — http://www.unimib.it/BEA